CLINICAL TRIAL: NCT03866434
Title: A Phase 1, Open-label, Single-sequence, Non-randomized, Crossover, Drug-Drug Interaction Study to Evaluate the Effect of Omeprazole on the Pharmacokinetics of SPD422 (Anagrelide Hydrochloride) in Healthy Adult Subjects
Brief Title: Study to Evaluate the Effect of Omeprazole on the Pharmacokinetics of SPD422 (Anagrelide Hydrochloride) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD422-113
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Results first posted 2020-04-24 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — anagrelide; Omeprazole

STUDY DESIGN:
Intervention Model Description: Single sequence crossover drug-drug interaction study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SPD422 + Omeprazole (Experimental): Participants will receive 1 milligram (mg) of SPD422 (Anagrelide hydrochloride) (2*0.5 mg) capsule orally on Day 1 in fasted state (10 hours prior to and until 4 hours following administration of anagrelide), followed by 40 mg of Omeprazole capsule orally once daily (prior to breakfast) on Days 2 to Day 7, followed by 1 mg of Anagrelide in fasted state in combination with Omeprazole 40 mg on Day 8.
  Interventions: Drug: SPD422; Drug: Omeprazole

INTERVENTIONS:
Drug: SPD422 — Participants will receive 1 mg of SPD422 (2*0.5 mg) capsule orally on Day 1 and 8 in fasted state.
  Other Names: Anagrelide hydrochloride
Drug: Omeprazole — Participants will receive 40 mg of Omeprazole orally once daily on Days 2 - 8.

SUMMARY:
This Phase 1, open-label, single-sequence, non-randomized, multiple-dose, crossover pharmacokinetic study is a single site study in the United States and will be conducted to assess the effect of a CYP1A2 inducer (omeprazole 40 mg once daily [QD]) on the pharmacokinetics of anagrelide (1 mg) when administered concurrently in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who has given, personally signed, and dated informed consent to participate in the study, in accordance with the International Conference on Harmonization Good Clinical Practice Guideline E6 (1996) and applicable regulations, before completing any study-related procedures.
* Age 18-45 years inclusive at the time of consent. The date of signing informed consent is defined as the beginning of the Screening Period. This inclusion criterion will be assessed only at the Screening Visit.
* Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential. A female of non-childbearing potential (defined as a female who is post-menopausal [amenorrhea for at least 12 consecutive months], has had a hysterectomy, bilateral tubal ligation, bilateral oophorectomy or bilateral salpingectomy.
* Satisfactory medical assessment with no clinically significant or relevant abnormal findings as determined by medical/surgical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory evaluation (hematology, biochemistry, thyroid function, and urinalysis) that are likely to interfere with the participant's participation or ability to complete the study as assessed by the investigator.
* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Body mass index (BMI) between 18.5 and 30.0 kilograms per square meter (kg/m^2) inclusive; assessed only at the screening visit.
* Able to swallow (multiple capsules or tablets at 1 time or consecutively at 1 time) all investigational product.
* Healthy as determined by the investigator on the basis of screening evaluations.

Exclusion Criteria:

* Current or recurrent disease or conditions (example: cardiovascular, renal, liver, gastrointestinal, malignancy or other conditions) that could affect the absorption, action, or disposition of either omeprazole or anagrelide or its metabolites, or could affect clinical assessments or clinical laboratory evaluations.
* Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the participant unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the investigational product or study procedures.
* Significant illness, as judged by the investigator, within the 2 weeks of administration of the first dose of investigational product.
* Use of any medication (including prescription, over-the-counter, herbal, multivitamin, oral contraceptives and other hormonal contraceptive treatments, or homeopathic preparations) within the 30 days prior to the first dose of study drug or during the study through Day 9 (occasional use of acetaminophen is allowed).
* Treatment with any known hepatic and/or P450 enzyme-altering agents, including CYP1A2 inducers or inhibitors within 30 days prior to the first dose of investigational product. This includes: Strong inhibitor- ciprofloxacin, enoxacin, fluvoxamine, and zafirlukast; Moderate inhibitor- methoxsalen, mexiletine, and oral contraceptives; Moderate inducer- phenytoin, rifampin, ritonavir, smoking, teriflunomide; Inducer- lansoprazole
* A history of any of the following medical conditions:

  1. History of previous bone marrow suppression.
  2. History of hypersensitivity to the investigational product.
  3. History of adverse hematologic reaction, (such as neutropenia, thrombocytopenia, anemia) to any drug.
  4. History of symptomatic or clinically meaningful orthostatic hypotension or syncope, as assessed by the investigator.
  5. History of controlled or uncontrolled hypertension or a systolic blood pressure greater than or equal to (>=) 140 millimeters of mercury (mmHg) or diastolic blood pressure >= 90 mmHg at the Screening Visit or Day -1.
  6. Participant has any history of seizure disorder.
  7. History or presence of known structural cardiac abnormalities, syncope, cardiac conduction problems (PR interval greater than (>) 220 milliseconds (ms), second or third-degree heart block, bundle branch block [except congenital right bundle branch block], or prolonged QTc interval) or exercise-related cardiac events.
  8. History of alcohol or other substance abuse within the last year.
* A participant's alcohol consumption that fulfils one of the following: (Note: One alcohol unit=1 beer [12 ounce {oz}]=1 wine [5 oz]=1 liquor [1.5 oz])

  1. Has consumed alcohol within 2 days prior to the first dose of investigational product.
  2. Male participants who consume more than 3 units of alcohol per day.
  3. Female participants who consume more than 2 units of alcohol per day.
* Positive screening test results for alcohol, drugs of abuse, or pregnancy (females of childbearing potential only) at the Screening Visit or Day -1.
* A positive human immunodeficiency virus (HIV) antibody screen, hepatitis B surface antigen (HBsAG) or hepatitis C virus antibody (HCV) screen.
* Use of tobacco in any form (smoking or chewing) or other nicotine-containing products in any form (gum, patch) within 30 days prior to the first dose of investigational product and during the in-house stay at the CRC.
* A positive urine cotinine test that is >= 50 Nano grams per milliliter (ng/mL) at either the Screening Visit or on Day -1.
* Routine consumption of more than 2 units of caffeine per day or participants who experience caffeine-withdrawal headaches or have a history of caffeine-withdrawal headaches. (One caffeine unit is contained in the following items: one 6-oz cup of coffee, two 12-oz cans of cola, one 12-oz cup of tea, and three 1-oz chocolate bars. Decaffeinated coffee, tea, or cola are not considered to contain caffeine.)
* Consumption of grapefruit, Seville oranges, and/or products containing these items within 7 days prior to the first dose of investigational product.
* Donation of blood or blood products (egg, plasma, or platelets) within 60 days prior to the first dose of investigational product.
* Known or suspected intolerance or hypersensitivity to the investigational products (anagrelide or omeprazole) or closely related compounds, or any of the stated ingredients.
* Within 30 days prior to the first dose of investigational product:

  1. Have used an investigational product (if elimination half-life is <6 days, otherwise 5 half-lives).
  2. Have been enrolled in a clinical study (including vaccine studies) that, in the Investigator's opinion, may impact this Shire-sponsored study.
* Prior screen failure, participation, or enrollment in this study.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- New Orleans Center for Clinical Research, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at single site in United States of America from 26 February 2019 to 10 April 2019.
Pre-assignment Details: A total of 20 participants were enrolled and completed the study.
Groups:
- SPD422 + Omeprazole: Participants received 1 milligram (mg) of SPD422 (Anagrelide hydrochloride) (2*0.5 mg) capsule orally on Day 1 under fasted state (10 hours prior to and until 4 hours following administration of anagrelide), followed by 40 mg of Omeprazole capsule orally once daily (prior to breakfast) on Day 2 to Day 7, followed by 1 mg of Anagrelide under fasted state in combination with Omeprazole 40 mg on Day 8.
Period: Overall Study
Arm/Group | SPD422 + Omeprazole
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who had taken at least 1 dose of investigational product (anagrelide or omeprazole) and had at least 1 post dose safety assessment.
Arm/Group | SPD422 + Omeprazole
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (7.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Anagrelide (SPD422)
Description: Cmax of Anagrelide (SPD422) on Day 1 and Day 8 was reported. For PK outcome measures the reporting groups were split based on administration of Anagrelide alone (Day 1) and Anagrelide in combination with Omeprazole (Day 8) to provide statistical comparison in this single arm study.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 8, 12 hours on Day 1 and Day 8, 24 hours on Day 8
Population: Pharmacokinetic (PK) set included all participants who received at least 1 dose of investigational product (anagrelide or omeprazole) and had at least 1 measurable post dose plasma concentration.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- SPD422 (Day 1): Participants received 1 milligram (mg) of SPD422 (Anagrelide hydrochloride) (2*0.5 mg) capsule orally on Day 1 under fasted state (10 hours prior to and until 4 hours following administration of anagrelide).
- SPD422 + Omeprazole (Day 8): Participants received 40 mg of Omeprazole capsule orally once daily (prior to breakfast) on Day 2 to Day 7, followed by received 1 mg of Anagrelide under fasted state in combination with Omeprazole 40 mg on Day 8.
Arm/Group | SPD422 (Day 1) | SPD422 + Omeprazole (Day 8)
Number analyzed (Participants) | 20 | 20
nanogram per milliliter (ng/mL) | 5.028 (3.0357) | 3.180 (1.6707)
Statistical Analysis 1: Comparison: SPD422 (Day 1) vs SPD422 + Omeprazole (Day 8); The means of the log-transformed pharmacokinetic parameters were compared between the two treatments (anagrelide with omeprazole [Day 8] versus anagrelide alone [Day 1]). In order to estimate the magnitude of the treatment regimen differences, the geometric mean ratio (i.e., the least squares (LS) mean difference in the log-transformed parameters back transformed to the original scale) and their 90 percent (%) confidence intervals (CI) were calculated; Test type: Equivalence — 90% CIs of geometric mean ratios being within 80% to 125%; ANOVA; A 2-factor analysis of variance (ANOVA) model with fixed factors for treatment and participant was fitted to the natural logtransformed PK parameters; % ratio of Geometric LSmeans = 64.225, 90% CI 2-sided [53.212 to 77.516] — This analysis was performed based on the ratio of geometric LS means and 90% confidence interval for ratio of geometric means expressed as percent

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of 3-Hydroxy (OH)-Anagrelide (Active Metabolite of Anagrelide)
Description: Cmax of 3-OH-Anagrelide (Active Metabolite of Anagrelide) on Day 1 and Day 8 was reported. For PK outcome measures the reporting groups were split based on administration of Anagrelide alone (Day 1) and Anagrelide in combination with Omeprazole (Day 8) to provide statistical comparison in this single arm study.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 8, 12 hours on Day 1 and Day 8, 24 hours on Day 8
Population: PK set included all participants who received at least 1 dose of investigational product (anagrelide or omeprazole) and had at least 1 measurable post dose plasma concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SPD422 (Day 1) | SPD422 + Omeprazole (Day 8)
Number analyzed (Participants) | 20 | 20
ng/mL | 10.30 (3.9633) | 8.341 (2.7448)
Statistical Analysis 1: Comparison: SPD422 (Day 1) vs SPD422 + Omeprazole (Day 8); The means of the log-transformed pharmacokinetic parameters were compared between the two treatments (anagrelide with omeprazole [Day 8] versus anagrelide alone [Day 1]). In order to estimate the magnitude of the treatment regimen differences, the geometric mean ratio (i.e., the LS mean difference in the log-transformed parameters back transformed to the original scale) and their 90% CI were calculated; Test type: Equivalence — 90% CIs of geometric mean ratios being within 80% to 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; %ratio of Geometric LeastSquare(LS)means = 82.203, 90% CI 2-sided [71.501 to 94.507] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Zero to Last Time Point (AUC[0-t]) of Anagrelide (SPD422) in Plasma
Description: AUC(0-t) of Anagrelide (SPD422) in plasma on Day 1 and Day 8 was reported. For PK outcome measures the reporting groups were split based on administration of Anagrelide alone (Day 1) and Anagrelide in combination with Omeprazole (Day 8) to provide statistical comparison in this single arm study.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 8, 12 hours on Day 1 and Day 8, 24 hours on Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | SPD422 (Day 1) | SPD422 + Omeprazole (Day 8)
Number analyzed (Participants) | 20 | 20
hour*nanogram per milliliter (h*ng/mL) | 13.25 (5.9297) | 9.683 (4.6171)
Statistical Analysis 1: Comparison: SPD422 (Day 1) vs SPD422 + Omeprazole (Day 8); [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — 90% CIs of geometric mean ratios being within 80% to 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; % ratio of Geometric LS means = 73.705, 90% CI 2-sided [64.555 to 84.152] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Area Under the Concentration Versus Time Curve From Zero to Last Time Point (AUC[0-t]) of 3-Hydroxy (OH)-Anagrelide (Active Metabolite of Anagrelide) in Plasma
Description: AUC(0-t) of 3-OH-Anagrelide (Active Metabolite of Anagrelide) in Plasma on Day 1 and Day 8 was reported. For PK outcome measures the reporting groups were split based on administration of Anagrelide alone (Day 1) and Anagrelide in combination with Omeprazole (Day 8) to provide statistical comparison in this single arm study.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 8, 12 hours on Day 1 and Day 8, 24 hours on Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SPD422 (Day 1) | SPD422 + Omeprazole (Day 8)
Number analyzed (Participants) | 20 | 20
h*ng/mL | 39.51 (14.946) | 33.14 (10.816)
Statistical Analysis 1: Comparison: SPD422 (Day 1) vs SPD422 + Omeprazole (Day 8); [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — 90% CIs of geometric mean ratios being within 80% to 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; % ratio of Geometric LS means = 85.527, 90% CI 2-sided [78.163 to 93.584] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-infinity]) of Anagrelide (SPD422) in Plasma
Description: AUC(0-infinity) of Anagrelide (SPD422) in plasma on Day 1 and Day 8 was reported. For PK outcome measures the reporting groups were split based on administration of Anagrelide alone (Day 1) and Anagrelide in combination with Omeprazole (Day 8) to provide statistical comparison in this single arm study.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 8, 12 hours on Day 1 and Day 8, 24 hours on Day 8
Population: PK set included all participants who received at least 1 dose of investigational product (anagrelide or omeprazole) and had at least 1 measurable post dose plasma concentration. Here the number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SPD422 (Day 1) | SPD422 + Omeprazole (Day 8)
Number analyzed (Participants) | 20 | 17
h*ng/mL | 13.54 (5.9951) | 10.27 (4.6070)
Statistical Analysis 1: Comparison: SPD422 (Day 1) vs SPD422 + Omeprazole (Day 8); [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — 90% CIs of geometric mean ratios being within 80% to 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; % ratio of Geometric LS means = 73.007, 90% CI 2-sided [62.528 to 85.243] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-infinity]) of 3-Hydroxy (OH)-Anagrelide (Active Metabolite of Anagrelide) in Plasma
Description: AUC(0-infinity) of 3-OH-Anagrelide (Active Metabolite of Anagrelide) in Plasma on Day 1 and Day 8 was reported. For PK outcome measures the reporting groups were split based on administration of Anagrelide alone (Day 1) and Anagrelide in combination with Omeprazole (Day 8) to provide statistical comparison in this single arm study.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 8, 12 hours on Day 1 and Day 8, 24 hours on Day 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SPD422 (Day 1) | SPD422 + Omeprazole (Day 8)
Number analyzed (Participants) | 20 | 18
h*ng/mL | 40.85 (14.948) | 35.51 (11.190)
Statistical Analysis 1: Comparison: SPD422 (Day 1) vs SPD422 + Omeprazole (Day 8); [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — 90% CIs of geometric mean ratios being within 80% to 125%; ANOVA; [statistical method as in outcome 1, analysis 1]; % ratio of Geometric LS means = 86.504, 90% CI 2-sided [78.462 to 95.371] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily had a causal relationship with this treatment. An AE was considered a TEAE if it started on or after dosing on Day 1 or if it started before dosing on Day 1 but increased in severity on or after dosing on Day 1 through the end of the study. Number of participants with TEAEs and TESAEs were reported.
Time Frame: From start of study drug administration up to follow-up (up to Day 18)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SPD422 + Omeprazole
Number analyzed (Participants) | 20
Participants
  Treatment Emergent Adverse Events (TEAEs) | 9
  Treatment Emergent Serious Adverse Events (TESAEs) | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (up to Day 18)
Arm/Group | SPD422 + Omeprazole
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 9/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD422 + Omeprazole (N=20)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 7 (11)
Insomnia (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT03866434/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT03866434/SAP_001.pdf